CLINICAL TRIAL: NCT00255008
Title: SEASON South East Asian Study Of Novel Genotypes in Hepatitis C Infection: Pegylated-Interferon and Ribavirin Therapy (PEGATRON REDIPEN Combination Therapy (PEG-Intron® REDIPEN Plus REBETOL®)) in Treatment Naive Patients With Genotypes 1, 6, 7, 8, 9: A Comparison of Race and Genotype on Treatment Outcome.
Brief Title: Peg-Intron and Rebetol Therapy in Treatment of Naive Hepatitis C Patients: A Comparison of Race and Genotype on Treatment Outcome (Study P04212)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04212
Record Dates: First submitted 2005-11-15; First posted 2005-11-17 (Estimated); Results first posted 2010-01-06 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C, Chronic
Keywords: chronic hepatitis C; pegylated interferon alfa-2b; ribavirin; Asia
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Genotype 1 SEA PEG-IFN/RIB 48 w (Active Comparator): Genotype 1 hepatitis C virus (HCV)-infected Southeastern Asian (SEA) subjects treated for up to 48 weeks with PEG-Intron (peginterferon alfa-2b; PEG-IFN) REDIPEN and REBETOL (ribavirin; RIB) combination therapy
  Interventions: Biological: peginterferon alfa-2b; Drug: ribavirin
- Genotype 1 Caucasian PEG-IFN/RIB 48 w (Active Comparator): Genotype 1 HCV-infected Caucasian subjects treated for up to 48 weeks with PEG-Intron REDIPEN and REBETOL combination therapy
  Interventions: Biological: peginterferon alfa-2b; Drug: ribavirin
- Genotype 6, 7, 8, 9 SEA PEG-IFN/RIB 24 w (Experimental): Genotype 6, 7, 8, 9 HCV-infected SEA subjects randomized to treatment for 24 weeks with PEG-Intron REDIPEN and REBETOL combination therapy
  Interventions: Biological: peginterferon alfa-2b; Drug: ribavirin
- Genotype 6, 7, 8, 9 SEA PEG-IFN/RIB 48 w (Active Comparator): Genotype 6, 7, 8, 9 HCV-infected SEA subjects randomized to treatment for 48 weeks with PEG-Intron REDIPEN and REBETOL combination therapy
  Interventions: Biological: peginterferon alfa-2b; Drug: ribavirin

INTERVENTIONS:
Biological: peginterferon alfa-2b — Powder for injection in Redipen (50, 80, 100, 120, and 150 microgram strengths), subcutaneous, dose of 1.5 micrograms/kg, weekly for up to 48 weeks
  Other Names: SCH 54031, PegIntron REDIPEN
  Arms: Genotype 1 Caucasian PEG-IFN/RIB 48 w; Genotype 1 SEA PEG-IFN/RIB 48 w; Genotype 6, 7, 8, 9 SEA PEG-IFN/RIB 48 w
Drug: ribavirin — 200 mg capsules, oral, weight-based dose of 800, 1000, or 1200 mg daily for up to 48 weeks
  Other Names: SCH 18908, REBETOL
  Arms: Genotype 1 Caucasian PEG-IFN/RIB 48 w; Genotype 1 SEA PEG-IFN/RIB 48 w; Genotype 6, 7, 8, 9 SEA PEG-IFN/RIB 48 w
Biological: peginterferon alfa-2b — Powder for injection in Redipen (50, 80, 100, 120, and 150 microgram strengths), subcutaneous, dose of 1.5 micrograms/kg, weekly for up to 24 weeks
  Other Names: SCH 54031, PegIntron REDIPEN
  Arms: Genotype 6, 7, 8, 9 SEA PEG-IFN/RIB 24 w
Drug: ribavirin — 200 mg capsules, oral, weight-based dose of 800, 1000, or 1200 mg daily for up to 24 weeks
  Other Names: SCH 18908, REBETOL
  Arms: Genotype 6, 7, 8, 9 SEA PEG-IFN/RIB 24 w

SUMMARY:
This is a multicenter clinical trial designed to compare the efficacy of 48 weeks of therapy with pegylated (PEG)-Interferon/ribavirin in Southeastern Asian patients with genotype 1 chronic hepatitis C with 48 weeks of therapy with PEG-Interferon/ribavirin in Caucasian patients with genotype 1 chronic hepatitis C. This study is also designed to provide a randomized comparison of 24 weeks versus 48 weeks of therapy with PEG-Interferon/ribavirin in Southeastern Asian patients with genotypes 6-9. The primary endpoint is sustained virologic response, as defined by negative hepatitis C virus (HCV) ribonucleic acid (RNA) in serum at 24 weeks after therapy completion.

ELIGIBILITY:
Inclusion Criteria:

* Comply with all current Australian Schedule of Pharmaceutical Benefits S100 eligibility criteria.
* Able to give written informed consent and adhere to study visit schedule.
* South East Asian ethnicity (except for Caucasian Gt1/1b in comparator arm) i.e. born in Vietnam, Cambodia, Laos, Thailand, Hong Kong, and China or have both parents born in these countries.
* Genotype 1, 1a, 1b, 6, 6a, 6b, 7, 8, or 9, as classified by INNO-LiPA assay.
* Hemoglobin >=120 g/L (females), >=130 g/L (males).
* Platelet count >=100 x 10^9/L.
* Neutrophil count >=1.5 x 10^9/L.
* Negative pregnancy test for females.
* Thyroid stimulating hormone (TSH) within normal limits.

Exclusion Criteria:

* Participation in any other investigational drug program within 30 days of the Screening Visit.
* Human immunodeficiency virus (HIV) antibody positive or hepatitis B surface antigen (HBsAg) positive.
* Genotype 2, 3, 4, or 5, as classified by INNO-LiPA assay.
* Non South East Asian ethnicity (unless recruited to Caucasian GT1 comparator arm).
* Evidence of liver disease due to other disorders (e.g., hemachromatosis, Wilson's disease).
* Ongoing drug or alcohol abuse which in the opinion of the investigator would jeopardize the patient's ability to comply with study requirements.
* Inability to comply with study requirements for other reasons.
* Decompensated cirrhosis (Ascites, history of encephalopathy or bleeding varices, serum albumin <35 g/L, prothrombin time (PT) prolonged by greater than 3 sec).
* Present or prior history of severe psychiatric disease requiring hospitalization or medication.
* History of severe seizure disorder.
* History of autoimmune disorders (e.g., rheumatoid arthritis, inflammatory bowel disease, immune thrombocytopenic purpura, systemic lupus erythematosus, or other mixed connective tissue disease, psoriasis, optic neuritis).
* Poorly controlled thyroid disease.
* Creatinine clearance <50 mL/min.
* Severe cardiovascular disease.
* Hepatocellular cancer.
* Clinically significant ophthalmologic disorders.
* Hemoglobinopathies (e.g., thalassemia, sickle-cell anemia).
* Treatment or recent treatment with immunosuppressive agents (excluding short-term corticosteroid withdrawal), and immunosuppressed transplant recipients scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2005-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Genotype 1 SEA PEG-IFN/RIB 48 w: Genotype 1 hepatitis C virus (HCV)-infected Southeastern Asian (SEA) subjects treated for up to 48 weeks with PegIntron (peginterferon alfa-2b; PEG-IFN) REDIPEN and REBETOL (ribavirin; RIB) combination therapy
Period: Overall Study
Arm/Group | Genotype 1 SEA PEG-IFN/RIB 48 w | Genotype 1 Caucasian PEG-IFN/RIB 48 w | Genotype 6, 7, 8, 9 SEA PEG-IFN/RIB 24 w | Genotype 6, 7, 8, 9 SEA PEG-IFN/RIB 48 w
Started | 45 | 9 | 33 | 34
Completed | 13 (The study was terminated early and as a result only 42 patients completed the study.) | 0 | 17 | 12
Not Completed | 32 | 9 | 16 | 22
Not completed — Adverse Event | 1 | 1 | 2 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 2
Not completed — Did not meet viral reduction criteria | 4 | 5 | 0 | 1
Not completed — Withdrew consent | 0 | 0 | 2 | 0
Not completed — Sponsor request | 18 | 3 | 8 | 17
Not completed — Adverse lab experience | 1 | 0 | 0 | 0
Not completed — Other | 7 | 0 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Genotype 1 SEA PEG-IFN/RIB 48 w | Genotype 1 Caucasian PEG-IFN/RIB 48 w | Genotype 6, 7, 8, 9 SEA PEG-IFN/RIB 24 w | Genotype 6, 7, 8, 9 SEA PEG-IFN/RIB 48 w | Total
Number analyzed (Participants) | 45 | 9 | 33 | 34 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (11.06) | 43.6 (12.30) | 46.8 (10.56) | 46.3 (10.71) | 45.2 (10.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 4 | 15 | 12 | 50
  Male | 26 | 5 | 18 | 22 | 71

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Achieved a Sustained Virologic Response (SVR)
Description: SVR is defined as negative hepatitis C virus ribonucleic acid (HCV RNA) in serum at 24 weeks after therapy completion. The study was terminated early due to slow enrollment. The primary outcome measure could not be assessed.
Time Frame: 24 weeks after completion of either up to 24 or 48 weeks of therapy
Population: The study was terminated early due to slow enrollment. The primary outcome measure should be assessed with caution. No data was available at 24 weeks after therapy for the Genotype 1 Caucasian treatment group.
Measure: Number; unit: Participants
Arm/Group | Genotype 1 SEA PEG-IFN/RIB 48 w | Genotype 1 Caucasian PEG-IFN/RIB 48 w | Genotype 6, 7, 8, 9 SEA PEG-IFN/RIB 24 w | Genotype 6, 7, 8, 9 SEA PEG-IFN/RIB 48 w
Number analyzed (Participants) | 5 | 0 | 17 | 8
Participants | 4 |  | 13 | 7
Statistical Analysis 1: Comparison: Genotype 1 SEA PEG-IFN/RIB 48 w; Test type: Superiority or Other; Proportion of patients (%) = 80.0, 95% CI [28.36 to 99.49]
Statistical Analysis 2: Comparison: Genotype 6, 7, 8, 9 SEA PEG-IFN/RIB 24 w; Test type: Superiority or Other; Proportion of patients (%) = 76.47, 95% CI [50.10 to 93.19]
Statistical Analysis 3: Comparison: Genotype 6, 7, 8, 9 SEA PEG-IFN/RIB 48 w; Test type: Superiority or Other; Proportion of patients (%) = 87.50, 95% CI [47.35 to 99.48]

ADVERSE EVENTS:
Arm/Group | Genotype 1 SEA PEG-IFN/RIB 48w | Genotype 1 Caucasian PEG-IFN/RIB 48w | Genotype 6,7,8,9 SEA PEG-IFN/RIB 24w | Genotype 6,7,8,9 SEA PEG-IFN/RIB 48w
Serious Adverse Events (participants affected / at risk) | 2/45 | 0/9 | 3/33 | 1/34
Other Adverse Events (participants affected / at risk) | 42/45 | 9/9 | 32/33 | 32/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Genotype 1 SEA PEG-IFN/RIB 48w (N=45) | Genotype 1 Caucasian PEG-IFN/RIB 48w (N=9) | Genotype 6,7,8,9 SEA PEG-IFN/RIB 24w (N=33) | Genotype 6,7,8,9 SEA PEG-IFN/RIB 48w (N=34)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TOOTH ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COLLAPSE OF LUNG (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Genotype 1 SEA PEG-IFN/RIB 48w (N=45) | Genotype 1 Caucasian PEG-IFN/RIB 48w (N=9) | Genotype 6,7,8,9 SEA PEG-IFN/RIB 24w (N=33) | Genotype 6,7,8,9 SEA PEG-IFN/RIB 48w (N=34)
ANAEMIA (Blood and lymphatic system disorders) | 6 (7) | 1 (1) | 0 (0) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (4) | 0 (0) | 2 (2) | 0 (0)
EAR DISORDER (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
TINNITUS (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERTHYROIDISM (Endocrine disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
DRY EYE (Eye disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
VISION BLURRED (Eye disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 5 (5) | 2 (3) | 5 (6) | 8 (9)
DRY MOUTH (Gastrointestinal disorders) | 3 (3) | 0 (0) | 7 (7) | 7 (7)
DYSPEPSIA (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 1 (2) | 0 (0) | 2 (2) | 0 (0)
MOUTH ULCERATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
NAUSEA (Gastrointestinal disorders) | 5 (6) | 4 (4) | 9 (10) | 11 (11)
ORAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
AXILLARY PAIN (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHILLS (General disorders) | 1 (1) | 2 (4) | 1 (2) | 2 (2)
FATIGUE (General disorders) | 16 (17) | 8 (8) | 12 (12) | 11 (11)
FEELING COLD (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
INFLUENZA LIKE ILLNESS (General disorders) | 13 (13) | 5 (5) | 20 (21) | 16 (17)
INJECTION SITE ERYTHEMA (General disorders) | 7 (7) | 3 (3) | 9 (9) | 11 (11)
INJECTION SITE RASH (General disorders) | 4 (5) | 0 (0) | 1 (1) | 3 (3)
INJECTION SITE REACTION (General disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
IRRITABILITY (General disorders) | 3 (3) | 4 (4) | 6 (6) | 3 (3)
MALAISE (General disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 13 (13) | 0 (0) | 5 (5) | 7 (7)
THIRST (General disorders) | 3 (3) | 0 (0) | 2 (2) | 2 (2)
ULCER (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SEASONAL ALLERGY (Immune system disorders) | 2 (2) | 0 (0) | 3 (3) | 3 (3)
HERPES SIMPLEX (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
HAEMOGLOBIN DECREASED (Investigations) | 4 (5) | 1 (1) | 2 (2) | 5 (5)
LYMPH NODE PALPABLE (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
WEIGHT DECREASED (Investigations) | 9 (9) | 0 (0) | 0 (0) | 1 (1)
ANOREXIA (Metabolism and nutrition disorders) | 6 (6) | 1 (1) | 0 (0) | 3 (3)
DECREASED APPETITE (Metabolism and nutrition disorders) | 12 (13) | 7 (7) | 14 (14) | 17 (17)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 7 (7) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 7 (7) | 1 (1)
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 8 (10) | 4 (4) | 11 (11) | 11 (13)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 4 (4)
SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
AMNESIA (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) | 3 (3)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
DIZZINESS (Nervous system disorders) | 9 (11) | 3 (3) | 8 (8) | 13 (14)
DYSGEUSIA (Nervous system disorders) | 4 (4) | 2 (2) | 2 (2) | 1 (1)
HEADACHE (Nervous system disorders) | 9 (12) | 1 (1) | 14 (14) | 13 (14)
LETHARGY (Nervous system disorders) | 6 (6) | 0 (0) | 14 (17) | 13 (14)
AGITATION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
DEPRESSED MOOD (Psychiatric disorders) | 1 (1) | 4 (4) | 5 (5) | 2 (2)
DISORIENTATION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 14 (17) | 4 (5) | 16 (16) | 14 (15)
MOOD ALTERED (Psychiatric disorders) | 3 (3) | 0 (0) | 1 (1) | 3 (3)
MOOD SWINGS (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
SLEEP DISORDER (Psychiatric disorders) | 3 (3) | 1 (1) | 2 (2) | 4 (5)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GENITAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0) | 6 (6) | 4 (4)
DRY THROAT (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 2 (2) | 2 (2)
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 1 (1) | 3 (3)
ALOPECIA (Skin and subcutaneous tissue disorders) | 17 (17) | 2 (2) | 11 (11) | 17 (17)
DRY SKIN (Skin and subcutaneous tissue disorders) | 12 (13) | 6 (6) | 13 (13) | 11 (13)
PRURITUS (Skin and subcutaneous tissue disorders) | 13 (19) | 6 (6) | 11 (11) | 9 (9)
RASH (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 8 (10) | 8 (8)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
HERNIA REPAIR (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
PALLOR (Vascular disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less